CLINICAL TRIAL: NCT06551493
Title: The Assessment of Postnatal Perineal Wound: Perspectives of Midwives and Women.
Brief Title: Postnatal Perineal Wound Assessment
Status: Recruiting | Type: Observational
Sponsor: Oxford Brookes University (Other)
Responsible Party: Principal Investigator, Giada Giusmin, Senior Lecturer in Midwifery, Oxford Brookes University
Other Study IDs: 334946
Record Dates: First submitted 2024-08-08; First posted 2024-08-13 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2024-08

CONDITIONS: Perineum; Wound
MeSH Terms: conditions — Wounds and Injuries | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Postnatal women
  Interventions: Other: Observation of postnatal wound assessment; Other: Interview
- Registered midwives
  Interventions: Other: Observation of postnatal wound assessment; Other: Interview

INTERVENTIONS:
Other: Observation of postnatal wound assessment — Observation of postnatal wound assessment
Other: Interview — Interview to elicit individual perspectives of wound assessment

SUMMARY:
Around 85% of women who give birth vaginally experience a perineal wound, which could be a tear or an incision between the vaginal opening and the anus. Despite that, there is often insufficient exploration of how postnatal perineal wound assessment is conducted in healthcare research.

Clinical guidelines from the National Institute for Health and Care Excellence (NICE) touch on the typical signs of wound infection but do not offer detailed guidance on the execution of perineal assessment. Existing research evidence is mostly focused on long-term complications, management of perineal trauma immediately after birth or severe perineal trauma. The limited research on perineal wound care highlights how poor communication and information provision harm women at a physical and psychological level, negatively affecting daily tasks such as caring for their newborns.

Although there have been few studies examining women's or midwives' perspectives on perineal wound assessment in the context of uncomplicated wounds, their perspectives have never been jointly investigated to produce a comprehensive overview. Moreover, no research has had a clinical focus, investigating how the assessment is conducted in practice and what informs this practice, except from women's reports of perceived sub-standard care received.

Therefore, this proposed research is clinically grounded and aims to explore women's and midwives' perspectives on postnatal perineal wound assessment. This is needed to identify evidence-based practices, or lack thereof, in order to determine ways in which the experience can be improved for women and to have a more positive impact on their wellbeing.

Eight to ten pairs of midwives-women will be first observed whilst the routine assessment is conducted to understand what happens during this episode of care, and then they will be separately interviewed within a few days to gather further understanding. Recruitment will be in a single centre, which is a tertiary unit in the UK.

ELIGIBILITY:
Inclusion Criteria:

Midwives:

* NMC Registered midwives
* Working in the NHS
* Working in the community or postnatal ward
* Who assess perineal wounds

Women:

* Postnatal women who had a vaginal birth within the last ten days and had an uncomplicated perineal tear (first, second-degree or episiotomy).
* Had a healthy newborn (for example, the newborn is not currently admitted to newborn intensive care or the woman did not have a stillbirth)
* Located in the community or in hospital being cared for by midwives, within ten days postpartum when postnatal perineal wound assessment occurs.
* Over the age of 18, who can consent to participation
* English-speaking

Exclusion Criteria:

Midwives:

* Non-registered midwives and those working outside the NHS
* Who do not perform postnatal perineal wound assessment due to clinical settings or task restrictions.

Women:

* Who had a cesarean section
* Who had a stillbirth or fetal/neonatal complications
* Who had a vaginal birth but sustained severe perineal tears (third or fourth-degree tears)
* Who have not received NHS care or are outside standard postnatal locations
* Who are over 10 days postpartum at the time of perineal wound assessment
* Who are below the age of 18
* Non-English-speaking women

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Midwives and postnatal women
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Survey. How midwives conduct postnatal perineal wound assessment step-by-step. | 10 days postnatal
Survey women's experiences of postnatal perineal wound assessment, i.e. emotional or physical discomfort. | 10 days postnatal

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford University Hospital NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided